CLINICAL TRIAL: NCT02392520
Title: GnRH Antagonist in the Luteal Phase Compared to Conventional Treatment in Women With Severe Early Ovarian Hyperstimulation Syndrome (OHSS) in Whom All Embryos Are Cryopreserved
Brief Title: Luteal Antagonist Versus Conventional Treatment in Women With Severe Early Ovarian Hyperstimulation Syndrome (OHSS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eugonia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: luteal antag OHSS RCT
Record Dates: First submitted 2015-03-13; First posted 2015-03-19 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Ovarian Hyperstimulation Syndrome
Keywords: severe OHSS; antagonist administration; conventional treatment
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome | interventions — cetrorelix; LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antagonist (Experimental): 0.25 mg GnRH antagonist cetrorelix will be administered once daily for 4 days, starting on the day of severe early OHSS diagnosis
  Interventions: Drug: cetrorelix (cetrotide)
- Conventional (Placebo Comparator): Women with severe early OHSS will be treated with conventional treatment, such as intravenous albumin administration, paracentesis of ascitic fluid, either on an outpatient or inpatient basis.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: cetrorelix (cetrotide) — 0.25 mg GnRH antagonist cetrorelix will be administered once daily for 4 days, starting on the day of severe early OHSS diagnosis
  Other Names: GnRH antagonist
  Arms: Antagonist
Drug: Placebo — intravenous albumin administration, paracentesis of ascitic fluid, correction of electrolyte imbalance and intravascular volume
  Other Names: conventional treatment
  Arms: Conventional

SUMMARY:
The study aims to compare the novel method of GnRH antagonist administration in the luteal phase versus conventional treatment in IVF patients who develop severe early ovarian hyperstimulation syndrome and have all their embryos cryopreserved.

DETAILED DESCRIPTION:
GnRH antagonist administration in the luteal phase has been proposed as a strategy for the treatment of established severe early OHSS, causing rapid regression of the syndrome on an outpatient basis. The approach has been described as tertiary OHSS prevention, thereby complementing the primary prevention (GnRH antagonist protocol) and secondary prevention (GnRH agonist trigger) that constitute the OHSS-free clinic concept. No randomized controlled trials (RCT) exist to date comparing luteal GnRH antagonist administration versus conventional treatment.

The aim of the present study is to compare the novel method of GnRH antagonist administration in the luteal phase versus conventional treatment with primary outcome time to severe OHSS regression, in IVF patients who develop severe early OHSS and have all their embryos cryopreserved.

ELIGIBILITY:
Inclusion Criteria:

* Women with established severe early OHSS.
* Criteria for the diagnosis of severe OHSS require:

  * the presence of moderate (or higher) ascites and at least two of the following:

    * enlarged ovaries (>100 mm maximal diameter),
    * haematocrit (Ht) >45%,
    * white blood cell count (WBC) >15,000/mm3.

Exclusion Criteria:

* Women not fulfilling the above criteria

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-03 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Time to severe OHSS regression | 2- 21 days after severe OHSS diagnosis

SECONDARY OUTCOMES:
Need for patient hospitalization | 2- 21 days after severe OHSS diagnosis
Hematocrit levels | 8 days after severe early OHSS diagnosis
White blood cells | 8 days after severe early OHSS diagnosis
Diameter of ovaries | 8 days after severe early OHSS diagnosis
Quantity of ascites | 8 days after severe early OHSS diagnosis
Estradiol levels | 8 days after severe early OHSS diagnosis
Progesterone levels | 8 days after severe early OHSS diagnosis
Serum levels of vascular endothelial growth factor (VEGF) | 8 days after severe early OHSS diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: George T Lainas, MD, Principal Investigator — Barts and The London NHS Trust (ART Unit)
Locations (1):
- Eugonia Unit of Assisted Reproduction, Athens, Greece

REFERENCES:
- [Background] Lainas TG, Sfontouris IA, Zorzovilis IZ, Petsas GK, Lainas GT, Kolibianakis EM. Management of severe early ovarian hyperstimulation syndrome by re-initiation of GnRH antagonist. Reprod Biomed Online. 2007 Oct;15(4):408-12. doi: 10.1016/s1472-6483(10)60366-5. PMID 17908403
- [Background] Lainas TG, Sfontouris IA, Zorzovilis IZ, Petsas GK, Lainas GT, Iliadis GS, Kolibianakis EM. Management of severe OHSS using GnRH antagonist and blastocyst cryopreservation in PCOS patients treated with long protocol. Reprod Biomed Online. 2009 Jan;18(1):15-20. doi: 10.1016/s1472-6483(10)60419-1. PMID 19146764
- [Background] Lainas TG, Sfontouris IA, Zorzovilis IZ, Petsas GK, Lainas GT, Alexopoulou E, Kolibianakis EM. Live births after management of severe OHSS by GnRH antagonist administration in the luteal phase. Reprod Biomed Online. 2009 Dec;19(6):789-95. doi: 10.1016/j.rbmo.2009.09.021. PMID 20031018
- [Background] Lainas GT, Kolibianakis EM, Sfontouris IA, Zorzovilis IZ, Petsas GK, Tarlatzi TB, Tarlatzis BC, Lainas TG. Outpatient management of severe early OHSS by administration of GnRH antagonist in the luteal phase: an observational cohort study. Reprod Biol Endocrinol. 2012 Aug 31;10:69. doi: 10.1186/1477-7827-10-69. PMID 22938051
- [Background] Lainas GT, Kolibianakis EM, Sfontouris IA, Zorzovilis IZ, Petsas GK, Lainas TG, Tarlatzis BC. Pregnancy and neonatal outcomes following luteal GnRH antagonist administration in patients with severe early OHSS. Hum Reprod. 2013 Jul;28(7):1929-42. doi: 10.1093/humrep/det114. Epub 2013 Apr 26. PMID 23624582
- [Background] Lainas GT, Kolibianakis EM, Sfontouris IA, Zorzovilis IZ, Petsas GK, Lainas TG, Tarlatzis BC. Serum vascular endothelial growth factor levels following luteal gonadotrophin-releasing hormone antagonist administration in women with severe early ovarian hyperstimulation syndrome. BJOG. 2014 Jun;121(7):848-55. doi: 10.1111/1471-0528.12572. Epub 2014 Feb 12. PMID 24621101